CLINICAL TRIAL: NCT00320502
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Determine the Effects of BXT-51072 on CK-MB in High-Risk Type 2 Diabetic Patients Undergoing Elective Percutaneous Coronary Intervention
Brief Title: A Phase 2 Study to Determine the Effects of BXT-51072 in Diabetic Patients Undergoing Angioplasty (PCI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synvista Therapeutics, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BXT-203
Record Dates: First submitted 2006-04-30; First posted 2006-05-03 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Acute Coronary Syndrome; Type 2 Diabetes
MeSH Terms: conditions — Acute Coronary Syndrome; Diabetes Mellitus, Type 2 | interventions — BXT 51072

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: BXT-51072

SUMMARY:
The purpose of this study is to determine the safety and feasibility of BXT-51072 as a cardioprotective agent in diabetics undergoing elective angioplasty / percutaneous intervention (PCI), a procedure to "open" coronary arteries.

BXT-51072 belongs to a class of drugs called "glutathione peroxidase mimics." BXT-51072 works by imitating a substance produced in various tissues in the body, which prevents damage of the heart and blood vessels.

DETAILED DESCRIPTION:
Following screening, baseline measurements and informed consent, patients will receive BXT-51072 40 mg or placebo in a 2:1 ratio, 30 minutes before their scheduled PCI and then three times per day for 2 days. There will be 5 treatment visits and 3 follow-up visits.

Blood samples will be obtained for CK-MB, troponin and routine chemistry. A 24-hour continuous electrocardiogram will be obtained following the PCI and regular electrocardiograms will be obtained during the study and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Scheduled for elective angioplasty with acute coronary syndrome within 72- hours or MI within 7 days

Exclusion Criteria:

* CK-MB above normal
* Elevated troponin not showing a decreasing value
* Congestive heart failure
* Atrial fibrillation or left bundle branch block
* Uncontrolled diabetes

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change in CK-MB
Safety

SECONDARY OUTCOMES:
Change in troponin
Myocardial ischemia by 24-hour continuous 12-lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Banai, MD, Principal Investigator — Sourasky Medical Center, Tel Aviv, Israel; Ariel Roguin, MD, PhD, Principal Investigator — Rambam Medical Center, Haifa, Israel
Locations (4):
- Israel (4):
  - Rambam Medical Center, Haifa
  - Western Galilee Hospital, Nahariya
  - Rivka Sieff Hospital, Safed
  - Sourasky Medical Center, Tel Aviv